CLINICAL TRIAL: NCT02298517
Title: Application of Breathing Exercises With Load Inspiratory Postoperative Abdominal Surgery: a Randomized Clinical Trial Blind
Brief Title: Application Breathing Exercises With Load Inspiratory Postoperative Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Eli Maria Pazzianotto Forti, PhD, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Carol2013; UnimepCarol2013 (Registry Identifier: UnimepCarol2013)
Record Dates: First submitted 2013-12-12; First posted 2014-11-24 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Pulmonary Atelectasis; Respiratory Tract Diseases; Pathological Conditions, Signs and Symptoms
Keywords: Morbid obesity; bariatric surgery; Respiratory muscle endurance; Respiratory muscle strength; spirometry; physiotherapy
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Tract Diseases; Pathological Conditions, Signs and Symptoms; Obesity, Morbid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (No Intervention): Individuals will be treated with conventional physiotherapy according to the routine service of physiotherapy of the hospital.
- Incentive spirometry to flow (Experimental): Was determined for this study that the flow of inspired air will be sufficient to raise up to three spheres. In addition to direct them to do explosive, fast and deep, lifting the ball explosively breaths. Every fifteen inspirations volunteers will be invited to rest for intervals of 30-60 seconds and repeat six times. The use of incentive spirometry was adapted from the recommendations of the American Association for Respiratory Care (1991).
  Interventions: Procedure: incentive spirometry
- incentive spirometry to volume (Experimental): Use of this incentive spirometry will be done as follows: the participants will be instructed to inhale deeply through the mouthpiece, to total lung capacity, starting from functional residual capacity. Will be performed 6 sets of 15 breaths each (deep, slow and sustained) intervals with 30-60 seconds between each series.
  Interventions: Procedure: incentive spirometry
- inspiratory load equipment-Threshold (Experimental): This group will use the device Threshold™. Where adjustment is considered 40% of PNSN achieved by the patient evaluation. The volunteer will be instructed to remain in a supine position with 45 ° fowler comfortably with arms and shoulders relaxed and perform an inspiration with enough force to overcome the linear load of the device, then make a normal expiration. This study was determined to carry six sets of 15 repetitions. The rest will be about one to two minutes in each intervention.
  Interventions: Procedure: inspiratory load equipment
- inspiratory load equipment-Power breathe (Experimental): To exercise inspiratory muscle in this group will be used device Power breathe ® K2 have the same resistance setting, allowing us to tailor your level of inspiratory muscles. Such adjustment will be made considering 40% of PNSN achieved by the patient in the assessment sniff. For its implementation, the patient will be lying with a tilt of the head of the litter at 45 °, the patient will be asked to inspire to overcome the resistance of the linear unit and after performing a normal expiration. This group will also be achieved 6 series with 15 repetitions each, with an interval of one to two minutes between sets.
  Interventions: Procedure: inspiratory load equipment

INTERVENTIONS:
Procedure: incentive spirometry — Incentive spirometry to flow and incentive spirometry to volume
  Arms: Incentive spirometry to flow; incentive spirometry to volume
Procedure: inspiratory load equipment — Threshold and Power breathe
  Arms: inspiratory load equipment-Power breathe; inspiratory load equipment-Threshold

SUMMARY:
The aim of this study is to evaluate the effects of the use of breathing exercises with inspiratory loading on respiratory muscle strength and endurance, lung volumes and capacities and thoracoabdominal mobility in patients after bariatric surgery.

It is believed that the use of inspiratory load may mitigate the negative effects of surgical trauma on respiratory muscle dysfunction, preserving respiratory muscle strength, lung volumes and diaphragm mobility, thus reducing the risk of pulmonary complications in the postoperative period.

DETAILED DESCRIPTION:
This is a prospective, randomized and blinded study, where volunteers will be selected anthropometric measurements, assessment of lung volumes and capacities, through spirometry, thoracoabdominal mobility through the circumference, assessment of inspiratory muscle strength and endurance.

After these evaluations will be done by lottery randomization, where the volunteers will be divided into five groups. They are: control, incentive spirometry to flow, the volume incentive spirometry, Threshold ™, Power breathe ®, according to their resources to be performed during the postoperative period. Each appeal will be held in 6 sets of 15 repetitions, totaling seven sessions, two in the immediate postoperative period, and five on the first postoperative day. At the end of the intervention volunteers will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 40 and 55 Kg/m²
* Aged between 25 and 55 years
* Submitted to Roux-en-Y type gastric by-pass by laparotomy
* Normal preoperative pulmonary function test

Exclusion Criteria:

* Hemodynamic instability
* Hospital stay longer than three days
* Presence of postoperative complications
* Smoking

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
EVALUATION OF INSPIRATORY MUSCLE ENDURANCE | Preoperatively and on the high hostitalar - On day 1 and day 3
  The endurance test is performed using the Power breathe ® K3.
  According to Basso and Costa (2012), this assessment divided into two tests:
  * Test incremental: starting with 10 centimeters of water, the volunteer is instructed to breathe normally for two minutes, thereafter a further minute, the next two minutes of exercise load will be increased, and so on until the volunteer fails to reach the predetermined pressure for three consecutive breaths or present dyspnea and / or fatigue. The largest load that is sustained for at least one minute will be considered the value of sustained maximal inspiratory pressure (PImáxS).
  * Test constant: is conducted PImáxS to 80%, which is obtained in the previous test, and determined the time limit (Tlim) run 30 minutes. The stopping criteria are the same as the incremental test.

SECONDARY OUTCOMES:
EVALUATION OF LUNG VOLUMES AND CAPACITIES | Preoperatively and on the high hostitalar - On day 1 and day 3
  Spirometry was carried out according to the guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS) (2005). Three types of maneuver were used in order to evaluate the lung volumes and flows: Slow Vital Capacity (SVC), Forced Vital Capacity (FVC) and Maximum Voluntary Ventilation (MVV). The maneuvers were carried out until three acceptable and reproducible curves were obtained, not exceeding more than eight attempts. The values extracted from each maneuver were selected according to Pereira (2002), and the predicted values calculated using the equation proposed by Pereira et al. (1992) for Brazilians.

OTHER OUTCOMES:
THORACOABDOMINAL MOBILITY | Preoperatively and on the high hostitalar - On day 1 and day 3
  The measurement of thoracoabdominal mobility was performed by using a tape scaled in centimeters. In the standing position, the measurements were made at levels axillary, xiphoid and abdominal during rest, and at maximal inspiration and maximal expiration. At each level, the measurements were performed three times. It computed the highest value of inspiration and the lowest of expiration. The absolute difference between these values was considered the thoracoabdominal mobility.
EVALUATION OF MUSCLE STRENGTH INSPIRATORY | Preoperatively and on the high hostitalar - On day 1 and day 3
  The Sniff is an alternative non-invasive technique for the assessment of inspiratory muscle strength by sniff nasal inspiratory pressure (PNSN). The measurement is performed using a peak pressure generated by nasal nostril during a maximal sniff from functional residual capacity (FRC).
  The measurement will be performed with one nostril occluded by a silicone nasal plug, which remained connected to the digital manometer by a catheter approximately 1mm diameter (RUPPEL, 1994). The maneuver is a maximal sniff, with the mouth closed, from functional residual capacity (FRC). The Sniff Test will be held in ten maneuvers, with an interval of 30 seconds between each maneuver, being used as a selection criterion Sniff acceptable to generate a peak pressure regularly and a duration between 0 and 5 sec.

CONTACTS AND LOCATIONS:
Overall Officials: Eli M Pazzianotto-Forti, PhD, Principal Investigator — Universidade Metodista de Piracicaba
Locations (1):
- Universidade Metodista de Piracicaba (UNIMEP) 13400911, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Derived] Pazzianotto-Forti EM, da Costa Munno CM, Merino DFB, Simoes da Rocha MR, de Mori TA, Junior IR. Effects of Inspiratory Exercise With Linear and Nonlinear Load on Respiratory Variables Post-Bariatric Surgery. Respir Care. 2019 Dec;64(12):1516-1522. doi: 10.4187/respcare.05841. Epub 2019 Aug 6. PMID 31387894